CLINICAL TRIAL: NCT06671652
Title: Adaptation and Implementation of a Cherokee-based Participatory Research Project to Reduce CVD Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Melissa Lewis, Associate Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2097784
Record Dates: First submitted 2023-12-19; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will take part in a community building program in which Cherokee cultural, linguistic, and historical experts will met with the self-selected community groups approximately 1 x month for 5 months. Participants will complete homework assignments for each meeting and will complete a final presentation on the history and culture of their families and communities.
  Interventions: Behavioral: Duyugoda igalenisodi (Starting again the right way)

INTERVENTIONS:
Behavioral: Duyugoda igalenisodi (Starting again the right way) — Participants in the intervention arm will receive training and resources to build community resources and programming

SUMMARY:
This is a two phase project. Phase I is an online convenience sample to collect health and preference data for the intervention phase, as well as a partnership with community to co-create an intervention; Phase II. Phase II is an intervention to improve community connection and historical knowledge within Cherokee communities within the Cherokee Nation reservation involving consultation with Cherokee cultural and historical experts.

DETAILED DESCRIPTION:
1. Identify necessary program enhancements to maximize reach and acceptability of the intervention for primary prevention of CVD in Cherokee Nation adults. The new intervention will have a broad reach, and thus, potentially greater public health impact. By building on the well-established and popular intervention, RTR, the goal is to maximize the likelihood that this intervention will be culturally acceptable, logistically feasible, and financially sustainable.
2. Conduct a pilot study (n = 40) to demonstrate acceptability and feasibility of the adapted intervention and research methods. The expectation is that the intervention will be culturally acceptable to participants, and retention and data collection protocols will support feasibility of a larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Citizen of Cherokee tribe

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Pre; Post (study completion; within 6 months)
  Systolic and Diastolic

SECONDARY OUTCOMES:
Positive Mental Health Scale | Pre; Post (study completion; within 6 months)
  [1-6], Higher scores = better outcome
"Cultural Efficacy" | Pre; Post (study completion; within 6 months)
  [1-5], Higher scores indicate better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Lewis, Principal Investigator — University of Missouri School of Medicine
Locations (1):
- Cherokee Nation, Tahlequah, Oklahoma, United States